CLINICAL TRIAL: NCT00240799
Title: A Randomized, Double-Blind, Placebo-Controlled Study Evaluating Acetaminophen Extended Release (3900 mg/Day) in the Treatment of Osteoarthritis of the Hip or Knee.
Brief Title: An Effectiveness and Safety Study of Acetaminophen Extended Release Caplets in the Treatment of Osteoarthritis of the Hip or Knee.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002488
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis hip; osteoarthritis knee; acetaminophen
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip; Osteoarthritis, Knee

ARMS (2):
- 001 (Experimental): acetaminophen extended release
  Interventions: Drug: acetaminophen extended release
- 002 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: acetaminophen extended release
  Arms: 001
Drug: placebo
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate acetaminophen extended release (3900 mg/day) compared to placebo for safety and effectiveness in the relief of signs and symptoms of osteoarthritis of the hip or knee over 12 weeks

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled study to evaluate acetaminophen extended release 3900 mg/day compared with placebo in the relief of signs and symptoms of osteoarthritis of the hip or knee over 12 weeks. The hypothesis is that 3900 mg/day acetaminophen extended release is superior to placebo in the relief of signs and symptoms of osteoarthritis of the hip or knee with respect to the three primary effectiveness endpoints. Propoxyphene Hydrochloride Capsules, 65 mg, are used as rescue medication if subjects experience inadequate pain relief. The primary efficacy assessments are the average change from baseline through Week 12 for the WOMAC pain subscale score and the WOMAC physical function subscale score, and the subject's average global assessment of their response to therapy through Week 12. Safety assessments at study visits consist of monitoring adverse events, vital signs, study joint assessments and clinical laboratory determinations. Treatment consists of two acetaminophen 650 mg extended release caplets or two placebo caplets, administered orally every 8 hours for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of osteoarthritis of the hip or knee for a minimum of six months
* History of hip or knee pain due to osteoarthritis requiring the use of NSAIDs, acetaminophen or another analgesic agent on a regular basis (>= three days/week) for at least three months before the screening visit
* History of positive benefit with acetaminophen use for osteoarthritis pain
* History (ie, at any time in the past since diagnosis) of osteoarthritis pain of the hip or knee when not taking osteoarthritis analgesic medication
* Subjects must report a history of a pain level of moderate, moderately severe, or severe, a WOMAC pain score >= 65 at baseline, and a 20% or greater increase in their pain score relative to their score at screening

Exclusion Criteria:

* History of surgery, including arthroscopy, or major trauma to the study joint in the previous six months before the screening visit
* Grade 1 or grade 4 severity of the study joint based on the Kellgren and Lawrence radiographic criteria
* Signs of clinically important active inflammation of the study knee joint including redness, warmth, and/or a large, bulging effusion with the loss of normal contour at the screening and/or baseline visits
* Secondary osteoarthritis of the study joint including, but not limited to, septic arthritis, inflammatory joint disease, gout, Paget's disease of bone, articular fracture, major dysplasias or congenital abnormality, ochronosis, acromegaly, hemochromatosis, Wilson's disease, avascular necrosis, or primary osteochondromatosis
* History of acute inflammatory arthritis or pseudogout of the study joint.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Average change from baseline through Week 12 for WOMAC pain subscale score. Average change from baseline through Week 12 for WOMAC physical function subscale score. Subject's average global assessment of response to therapy through Week 12.

SECONDARY OUTCOMES:
Average change from baseline through Week 12 for: WOMAC stiffness subscale score; total WOMAC Osteoarthritis Index; and Nottingham Health Profile Energy subscale score

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- [Derived] Prior MJ, Harrison DD, Frustaci ME. A randomized, double-blind, placebo-controlled 12 week trial of acetaminophen extended release for the treatment of signs and symptoms of osteoarthritis. Curr Med Res Opin. 2014 Nov;30(11):2377-87. doi: 10.1185/03007995.2014.949646. Epub 2014 Aug 14. PMID 25121804
- [Derived] Kuffner EK, Temple AR, Cooper KM, Baggish JS, Parenti DL. Retrospective analysis of transient elevations in alanine aminotransferase during long-term treatment with acetaminophen in osteoarthritis clinical trials. Curr Med Res Opin. 2006 Nov;22(11):2137-48. doi: 10.1185/030079906x148346. PMID 17076974
- See also: An Effectiveness and Safety Study of Acetaminophen Extended Release Caplets in the Treatment of Osteoarthritis of the Hip or Knee — http://download.veritasmedicine.com/PDF/CR002488_CSR.pdf